CLINICAL TRIAL: NCT01364181
Title: The Impact of Udenafil on Exercise Capacity in Severe COPD Patients
Brief Title: The Impact of Udenafil on Exercise Capacity in Severe Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A PharmTech Co., Ltd. (Industry)
Responsible Party: Ho Il Yoon, M.D. Ph.D., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Udenafil
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-05

CONDITIONS: Dyspnea; Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension
Keywords: Udenafil; Chronic obstructive pulmonary disease; pulmonary hypertension; Phosphodiesterase 5 inhibitors; Exercise; Dyspnea
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Motor Activity | interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Udenafil (Experimental): Udenafil 50mg qd po
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — Udenafil 50mg qd po
  Other Names: Zydena

SUMMARY:
Pulmonary hypertension (PH) is a serious complication of COPD which is associated with shorter survival, more frequent exacerbation, and increased use of health resources. There is no effective pharmacological treatment for COPD-associated PH. Therefore, the investigators wanted to evaluate the effect of udenafil, a phosphodiesterase- 5 (PDE-5) inhibitor, on exercise capacity of severe COPD patients.

DETAILED DESCRIPTION:
Study design

* prospective, single arm, open-label study
* Udenafil 50mg qd po for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD who showed post-bronchodilator forced expiratory volume in 1 second (FEV1) less than 50% of predicted value

Exclusion Criteria:

* Acute exacerbation within 4 weeks of the study entry
* Coronary heart disease
* History of adverse event on PDE-5 inhibitors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
change of 6-minute walk distance | 8 weeks

SECONDARY OUTCOMES:
change of mean pulmonary artery pressure | 8 weeks
  change of lung function, SGRQ score, Borg index, oxygen saturation, mean pulmonary artery pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ho Il Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Park JS, Lim HJ, Cho YJ, Lee JH, Yoon HI, Lee CT. Udenafil improves exercise capacity in patients with chronic obstructive pulmonary disease: a prospective study. COPD. 2012 Aug;9(5):499-504. doi: 10.3109/15412555.2012.694922. Epub 2012 Sep 4. PMID 22946546